CLINICAL TRIAL: NCT04981574
Title: Comparison of the Effectiveness of the Thoracic Thrust Manipulation in People With Neck or Low Back Pain
Brief Title: Effectiveness Comparison of Thoracic Thrust Manipulation in People With Neck or Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Principal investigator, University of Jaén
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alcalá
Record Dates: First submitted 2021-07-07; First posted 2021-07-29 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Neck Pain; Low Back Pain
Keywords: neck pain; low back pain; spinal manipulation; acute pain
MeSH Terms: conditions — Neck Pain; Low Back Pain; Acute Pain | interventions — Massage

STUDY DESIGN:
Intervention Model Description: It is a controlled clinical trial with parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group: neck pain (Experimental)
  Interventions: Other: Massage and stretching on neck area and thoracic thrust manipulation
- B group: low back pain (Experimental)
  Interventions: Other: Massage and stretching on low back area and thoracic thrust manipulation

INTERVENTIONS:
Other: Massage and stretching on neck area and thoracic thrust manipulation — 1. Twenty (20) minutes massage in the neck area. The volunteer will be in prone position during the massage.
  2. Technical thrust manipulation in thoracic area. For this technique the volunteer will be in supine position with their arms folded on the chest (making a "V"). The therapist will locate one hand on the spinous processes to be treated, and the other one on the arms of the patient to make easier the manipulation.
  3. Ten (10) minutes specific stretching for the neck area. These stretching exercises shall be repeated twice a week by each volunteer. Stretching will be made on the trapezius superior, musculus levator scapulae and sternocleidomastoideus holding the position thirty (30) seconds. Each muscle stretch shall be repeated three times.
  Arms: A group: neck pain
Other: Massage and stretching on low back area and thoracic thrust manipulation — 1. Twenty (20) minutes massage in the low back area. The volunteer will be in prone position during the massage.
  2. Technical thrust manipulation in thoracic area. For this technique the volunteer will be in supine position with their arms folded on the chest (making a "V"). The therapist will locate one hand on the spinous processes to be treated, and the other one on the arms of the patient to make easier the manipulation.
  3. Ten (10) minutes specific stretching for the low back area. These stretching exercises shall be repeated twice a week by each volunteer. Stretching activities will be: cat-cow pose, lower back stretches and knee twist holding the position thirty (30) seconds. Each muscle stretch shall be repeated three times.
  Arms: B group: low back pain

SUMMARY:
Objective:

To compare the effectiveness of thoracic thrust manipulation, together with massages techniques and stretching, between people with neck pain versus people with low back pain.

Methods:

The research will be performed from August 2021 to October 2021 at the University of Alcala de Henares. (Madrid)

A minimum of forty-six (46) volunteers will participate in this research, and they will be divided in two groups of twenty-three (23). One group will be formed by candidates suffering from neck pain (group A) and the other one by candidate with low back pain (group B).

Both groups will receive the same treatment and specific stretching exercises as applicable in accordance to the pain area, e.g.: group A will get the massage and the stretching exercises more suitable for the neck pain and group B the same but for the low back pain. Nevertheless both groups will receive the same technical thrust manipulation in thoracic area.

All these treatments will be applied of the volunteers at the University of Alcalá.

The treatment includes the following activities:

1. Twenty (20) minutes massage in the pain area, as applicable.
2. Technical thrust manipulation in thoracic area.
3. Ten (10) minutes stretching in accordance to the pain area treated. The stretching shall be repeated twice a week by each volunteer.

A total of six (6) sessions will be carried out during six (6) weeks, one session per week.

Pain, disability, kinesiophobia, HRQoL will be assessed as follow:

1. Before first session. (In this evaluation will be also analyzed demographic variables i.e.: height, weight, age, gender, academic level, smoker/no smoker)
2. Between third and fourth session.
3. After sixth session.
4. Four weeks after sixth session.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Non-specific neck/low back pain for the last three (3) months before the first session.

Exclusion Criteria:

* Previous surgery in the areas covered by this research (neck and/or low back)
* Red flags: Cancer or tumor, fracture...
* Scoliosis or osteoporosis
* Neck or low back pain with radiculopathy symptoms
* Central nervous system involvement
* Fear to manipulation
* Neck pain associated with whiplash injuries on the last six (6) months
* Pregnant women
* Not understand, write and speak Spanish fluently

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Change in Neck and Low Back Pain | Baseline, 3 weeks, 6 weeks, and 10 weeks after intervention commencement
  using a Visual Analogue Scale (VAS) from 0 to 10

SECONDARY OUTCOMES:
Change in Neck Pain related disability | Baseline, 3 weeks, 6 weeks, and 10 weeks after intervention commencement
  Using the Neck Disability Index (NID) Questionnaire
Change in Health related quality of life (HRQoL) | Baseline, 3 weeks, 6 weeks, and 10 weeks after intervention commencement
  Using the SF-12 Quality of Life Questionnaire
Change in kinesiophobia | Baseline, 3 weeks, 6 weeks, and 10 weeks after intervention commencement
  Using the fear avoidance beliefs (FAB) questionnaire
Change in Low Back Pain related disability | Baseline, 3 weeks, 6 weeks, and 10 weeks after intervention commencement
  Using the Oswestry Disability Index (ODI) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Achalandabaso, Study Director — University of Jaén
Locations (1):
- Alicia Masip, Alcalá de Henares, Madrid, Spain